CLINICAL TRIAL: NCT01854164
Title: An 8 Weeks, Randomized, Double-blind, Placebo-controlled Clinical Trial for Anti-diabetic Effects of Hydrolyzed Ginseng Extract
Brief Title: Efficacy and Safety of Hydrolyzed Ginseng Extract on Impaired Fasting Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Ilhwa-FG-001
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Hyperglycemia
Keywords: HGE, impaired fasting glucose, clinical trial
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HGE(hydrolyzed ginseng extract) (Experimental): HGE capsules(2cap/d, 960mg/d) for 8 weeks.
  Interventions: Dietary Supplement: HGE (hydrolyzed ginseng extract)
- Placebo (Placebo Comparator): Placebo for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: HGE (hydrolyzed ginseng extract)
  Arms: HGE(hydrolyzed ginseng extract)
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of hydrolyzed ginseng extract(HGE) on glycemic status in subjects with impaired fasting glucose(IFG).

DETAILED DESCRIPTION:
This study was a 8 weeks, randomized, double-blind, placebo-controlled trial. Twenty subjects were randomly divided into HGE or a placebo group. Fasting and postprandial glucose profiles during oral glucose tolerance test (OGTT) were assessed before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-70 years with fasting glucose 100~126 mg/dL

Exclusion Criteria:

* Abnormal lipid profile values
* Acute/chronic inflammation
* Treated with corticosteroid within past 4 weeks
* Cardiovascular disease
* Allergic or hypersensitive to any of the ingredients in the test products
* History of disease that could interfere with the test products or impede their absorption
* Participation in any other clinical trials within past 2 months
* Renal disease
* Abnormal hepatic function
* Under hypolipidemic drugs therapy within past 3 months
* Under antipsychotic drugs therapy within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* History of alcohol or substance abuse
* Pregnancy or breast feeding

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Changes of blood glucose during OGTT(oral glucose tolerance test) | 8 weeks
  Changes of fasting and postprandial glucose during OGTT were assessed before(baseline) and after the intervention.

SECONDARY OUTCOMES:
Changes of blood insulin during OGTT. | 8 weeks
  Changes of blood insulin during OGTT were assessed before(baseline) and after the intervention.
Changes of glycated albumin, fructosamine, and lipid profile | 8 weeks
  Changes of glycated albumin, fructosamine, and lipid profile were assessed before(baseline) and after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods, Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea